CLINICAL TRIAL: NCT02460744
Title: A Phase II Study of 2-weeks of Adjuvant Whole Breast/Chest Wall and/or Regional Nodal Radiotherapy in Patients With Breast Cancer
Brief Title: 2-weeks of Adjuvant Radiotherapy in Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Budhi Singh Yadav, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHRT
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; hypofractionation; radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm treatment with radiation (Experimental): Patients with breast cancer will be given adjuvant hypofractionated radiotherapy
  Interventions: Radiation: Hypofractionation

INTERVENTIONS:
Radiation: Hypofractionation — Radiation dose of 34Gy in 10 fractions over 2 weeks.

SUMMARY:
The investigators at PGIMER have been practicing hypofractionation radiotherapy with a dose of 35Gy/15#/3wks to the chest wall in post mastectomy and 40Gy/16#/3wks in breast conservation in breast cancer patients for the last 4 decades. It is also a routine practice in UK and few centers in Canada. Hypofractionation reduces treatment time to half while maintaining cosmesis and gives control rates equal to conventional fractionation. As breast cancer is a leading cancer in females and radiation therapy is an important part of its local management, hypofractionation help the radiation centers worldwide to meet the growing need for radiation in breast cancer, particularly in developing countries where resources are limited. It also reduces the financial burden on the patient and family.

In this study the investigators want to reduce the treatment duration from 3 weeks to 2 weeks. The study will include 20 patients with breast cancer post mastectomy or after breast conservative surgery to be treated with a radiotherapy dose of 34Gy in 10 fractions over 2 weeks. Patients will be assessed for acute radiation toxicity weekly during treatment and after one month of completion of treatment.

DETAILED DESCRIPTION:
Patients to be included in this study will be pre-operatively staged according to American Joint Committee on Cancer (AJCC) 7th edition, International Union against cancer ( which uses TNM staging ) as stage I , stage II of breast carcinoma. Twenty patients of histologically proven post lumpectomy/mastectomy cases of carcinoma breast suitable for radiotherapy will be enrolled in this study. Patients would be evaluated at the Department of Radiotherapy PGIMER, Chandigarh by doing a thorough clinical examination followed by routine investigations which will include hemogram, liver function tests, kidney function tests, chest X-ray. Patients will be treated by standard rectangular tangential fields.The study will include 20 patients with breast cancer post mastectomy or after breast conservative surgery to be treated with a radiotherapy dose of 34Gy in 10 fractions over 2 weeks followed by a boost of 10Gy/5#/1wk in cases with intact breast. Acute toxicity will be assessed using a RTOG grading system. This will be carried out weekly during radiotherapy and for 4 weeks after treatment. If symptoms persist the patients will be assessed weekly until their reaction settles to RTOG grade 1 or less (Annexure I).

Statistical analyses The principle end point of the study is an analysis of acute toxicities, cosmetic score analysis. Skin, subcutaneous toxicity and cosmetic assessment will be done before treatment and then in regular follow up of the study. Chi-square test will be used to compare radiation toxicity parameters. Descriptive statistics including mean and standard deviation will be obtained for all variables. p values of <0.05 will be taken as significant. All tests would be performed using SPSS (Statistical Package for the Social Sciences) v.12.0.

ELIGIBILITY:
Inclusion Criteria:

* invasive carcinoma of the breast
* breast conservation surgery or mastectomy (reconstruction allowed but not with implant. Tissue expanders with distant metal ports are allowed)
* axillary staging &/or dissection
* complete microscopic excision of primary tumour
* pT1-3 pN0-2 M0 disease
* written informed consent
* able to comply with follow up N.B. Concurrent trastuzumab and hormone therapy is allowed

Exclusion Criteria:

* past history of malignancy except (i) basal cell skin cancer and CIN cervix uteri or (ii) non-breast malignancy allowed if treated with curative intent and at least 5 years disease free
* contralateral breast cancer, including DCIS, irrespective of date of diagnosis
* breast reconstruction using implants
* concurrent cytotoxic chemotherapy (sequential neoadjuvant or adjuvant cytotoxic therapy allowed)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
acute skin and subcutaneous toxicity assessed using a RTOG grading system | 1 month
  Acute toxicity will be assessed using a RTOG grading system.

SECONDARY OUTCOMES:
Cosmetic score analysis using Harvard/NSABP/RTOG Breast Cosmesis Grading Scale | Base line, one month and 6 months after completion of radiation
  Cosmetic score analysis will be done using Harvard/NSABP/RTOG Breast Cosmesis Grading Scale

CONTACTS AND LOCATIONS:
Overall Officials: Budhi S Yadav, MD, Principal Investigator — PGIMER, Chandigarh, India
Locations (1):
- Dr Budhi Singh Yadav, Chandigarh, N/A = Not Applicable, India

REFERENCES:
- [Derived] Yadav BS, Sharma SC. A Phase 2 Study of 2 Weeks of Adjuvant Whole Breast/Chest Wall and/or Regional Nodal Radiation Therapy for Patients With Breast Cancer. Int J Radiat Oncol Biol Phys. 2018 Mar 15;100(4):874-881. doi: 10.1016/j.ijrobp.2017.12.015. Epub 2017 Dec 16. PMID 29485066